CLINICAL TRIAL: NCT07001657
Title: Analgesic Efficacy of Pectoral Nerve Block and Serratus Posterior Superior Intercostal Plane Block in Breast Cancer Surgery; Randomized Controlled Trial
Brief Title: Pectoral Nerve Block and Serratus Posterior Superior Intercostal Plane Block in Breast Cancer Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Antalya Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Nilgun Kavrut Ozturk, Professor MD, Antalya Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: AEAHYE001
Record Dates: First submitted 2025-05-16; First posted 2025-06-03 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Nerve Block
Keywords: pectoral nerve block; Breast Cancer Surgery; Serratus Posterior Superior Intercostal Plane Block; Postoperative Pain; Patient Controlled Analgesia
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SPSIP Block (Active Comparator): Patients in this group will receive an ultrasound-guided Serratus Posterior Superior Intercostal Plane (SPSIP) block with 30 mL of 0.25% bupivacaine hydrochloride injected into the fascial plane between the serratus posterior superior muscle and the third rib, 30 minutes before surgery.
  Interventions: Procedure: SPSIP Block
- PECS II Block (Active Comparator): Patients in this group will receive an ultrasound-guided PECS II block with 30 mL of 0.25% bupivacaine hydrochloride (20 mL between the pectoralis minor and serratus anterior muscles, and 10 mL between the pectoralis major and minor muscles), 30 minutes before breast cancer surgery.
  Interventions: Procedure: PECS II Block

INTERVENTIONS:
Procedure: SPSIP Block — Patients in this group will receive an ultrasound-guided Serratus Posterior Superior Intercostal Plane (SPSIP) block with 30 mL of 0.25% bupivacaine hydrochloride injected into the fascial plane between the serratus posterior superior muscle and the third rib, 30 minutes before surgery.
  Arms: SPSIP Block
Procedure: PECS II Block — Patients in this group will receive an ultrasound-guided PECS II block with 30 mL of 0.25% bupivacaine hydrochloride (20 mL between the pectoralis minor and serratus anterior muscles, and 10 mL between the pectoralis major and minor muscles), 30 minutes before breast cancer surgery.
  Arms: PECS II Block

SUMMARY:
This randomized clinical trial aims to evaluate and compare the analgesic efficacy of the Pectoral Nerve Block (PECS II) and the Serratus Posterior Superior Intercostal Plane (SPSIP) Block in patients undergoing breast cancer surgery. The primary outcome is total opioid consumption in the first 24 hours. Secondary outcomes include pain scores (VAS), block performance time, number of needle passes, postoperative recovery quality (QoR-15), time to first analgesic request, and complications (hematoma, pneumothorax, local anesthetic toxicity, vascular puncture, infection).

DETAILED DESCRIPTION:
Study Objective This research aims to obtain objective data to demonstrate the effectiveness of two regional block techniques in acute pain management. The primary objective is to compare the effects of Pectoral Nerve Block (PECS II) and Serratus Posterior Superior Intercostal Plane Block (SPSIP) on total opioid consumption within the first 24 hours and on Visual Analog Scale (VAS) scores in patients undergoing breast cancer surgery. Secondary outcomes include evaluating the impact of these blocks on intraoperative opioid requirement and postoperative recovery quality.

Materials and Methods This prospective, randomized clinical study will include voluntary female patients aged 18-65 years, classified as American Society of Anesthesiologists (ASA) physical status I-III, with a body mass index (BMI) <35 kg/m². All participants will be informed about the study protocol in detail, and written informed consent will be obtained prior to inclusion. Patients will receive instruction on the use of the VAS for pain assessment, where 0 denotes no pain and 10 denotes the worst imaginable pain.

Patients who meet the exclusion criteria will be withdrawn from the study. Participants will be randomly assigned to one of two groups using a computer-generated simple randomization method (https://www.randomizer.org). Randomization will be performed by a team member uninvolved in patient care, who will also prepare sealed opaque envelopes to conceal group allocation until shortly before block administration.

Study Groups and Block Procedures Group SPSIP will receive a unilateral SPSIP block, and Group PECS-II will receive a unilateral PECS II block. All patients will be monitored with electrocardiography, peripheral oxygen saturation (SpO₂), and non-invasive blood pressure prior to the block. Premedication with intravenous midazolam (0.02 mg/kg) will be administered.

SPSIP Block:

The Serratus Posterior Superior Intercostal Plane (SPSIP) block will be performed 30 minutes prior to surgery with the patient in a sitting position. After skin disinfection with chlorhexidine, the skin and subcutaneous tissues will be anesthetized using 2-4 mL of 1% lidocaine (Aritmal®, Osel Pharmaceuticals, Turkey). A linear ultrasound probe (Mindray Diagnostic Ultrasound System, Model DC-T6) will be positioned along the medial border of the scapula at the level of the second and third ribs on the surgical side.

Anatomical landmarks, including the trapezius, rhomboid major muscle (RMM), serratus posterior superior muscle (SPSM), and the second and third ribs will be identified. Using an in-plane approach, a 21G 0.8×100 mm echogenic insulated needle (Echoplex®+, Vygon SA, Écouen, France) will be inserted into the fascial plane between the third rib and the SPSM. Proper needle placement will be confirmed with the injection of 1-2 mL isotonic saline. Upon confirmation and negative aspiration, 30 mL of 0.25% bupivacaine hydrochloride (Buvasin®, Vem Pharmaceuticals, Turkey) will be administered.

The block performance time, defined as the duration from initial ultrasound probe contact with the skin to the final withdrawal of the needle following injection, will be recorded.

PECS II Block:

Patients will be placed in the supine position, and the PECS II block will be administered. Prior to all blocks, the skin will be disinfected with chlorhexidine, and the skin and subcutaneous tissue will be anesthetized using 2-4 mL of 1% lidocaine (Aritmal®, Osel Pharmaceuticals, Turkey). A linear ultrasound probe (Mindray Diagnostic Ultrasound System, Model DC-T6) will be used and positioned at the level of the third and fourth ribs along the mid-axillary line on the surgical side.

Key anatomical landmarks including the pectoralis major, pectoralis minor, and serratus anterior muscles, as well as the third and fourth ribs will be identified. Using an in-plane approach, a 21G 0.8×100 mm echogenic insulated needle (Echoplex®+, Vygon SA, Écouen, France) will be advanced into the fascial plane between the pectoralis minor and serratus anterior muscles. Proper needle placement will be confirmed by the injection of 1-2 mL of isotonic saline, followed by the administration of 20 mL of 0.25% bupivacaine hydrochloride (Buvasin®, Vem Pharmaceuticals, Turkey).

The needle will then be redirected to the fascial plane between the pectoralis major and pectoralis minor muscles. Following negative aspiration and confirmation of correct positioning with 1-2 mL of isotonic saline, 10 mL of 0.25% bupivacaine will be injected.

The block performance time defined as the time interval from the ultrasound probe's contact with the skin to the withdrawal of the needle after the final injection will be recorded.

General Anesthesia Upon entry into the operating room, patients will be monitored with electrocardiography, peripheral oxygen saturation (SpO₂), and non-invasive blood pressure. Anesthesia will be induced with intravenous propofol (2 mg/kg, Polifarma Pharmaceutical Industry and Trade Inc., Ergene, Turkey), fentanyl citrate (1.5 mcg/kg, Polifarma Pharmaceutical Industry and Trade Inc., Ergene, Turkey), and rocuronium bromide (0.6 mg/kg, Muscuron®, Koçak Farma Pharmaceutical and Chemical Industry Co., Turkey).

Anesthesia maintenance will be provided using 2% sevoflurane in a 50% oxygen-air mixture and a continuous remifentanil infusion at 0.05 mcg/kg/min. Mechanical ventilation settings will be adjusted to deliver a tidal volume of 6-8 mL/kg with end-tidal CO₂ maintained at 30-35 mmHg. Anesthetic depth will be monitored continuously using a Bispectral Index (BIS™) monitor (Medtronic plc, Dublin, Ireland), targeting a BIS value of 40-60. If heart rate or mean arterial pressure increases >20% from baseline, the remifentanil dose will be titrated accordingly.

Thirty minutes before the end of surgery, all patients will receive 15 mg/kg of intravenous paracetamol (e.g., Paracerol®, Polifarma Pharmaceutical Industry and Trade Inc., Ergene, Turkey) and 1 mg/kg of intravenous tramadol. To prevent nausea and vomiting, 0.15 mg/kg of intravenous ondansetron will be administered. Patients with adequate spontaneous ventilation will be extubated and transferred to the post-anesthesia care unit (PACU).

Hemodynamic Monitoring Heart rate, systolic blood pressure, diastolic blood pressure, mean arterial pressure, and oxygen saturation will be recorded at the following time points: pre-induction (baseline), 5 minutes after induction, 5 minutes after surgical incision, 15 minutes after incision, and at the end of surgery.

Postoperative Pain and Analgesic Use Pain will be assessed using the VAS at rest (static) and during movement (dynamic) at 1, 3, 6, 12, and 24 hours postoperatively. All patients will use patient-controlled analgesia (PCA) without a basal infusion. The PCA device will be set to deliver 1 mg of morphine (0.2 mg/mL concentration) with a 10-minute lockout interval. Patients will be instructed to press the PCA button when VAS ≥4. Intravenous paracetamol will be administered every 8 hours. Rescue analgesia with intravenous tramadol (1 mg/kg) will be provided if VAS scores remain ≥4. The total amounts of opioids, NSAIDs, and other analgesics will be recorded.

Postoperative Recovery Quality Postoperative recovery will be assessed using the 15-item Quality of Recovery-15 (QoR-15) questionnaire, which evaluates five domains: pain, physical comfort, physical independence, psychological support, and emotional state.

Patient and Surgeon Satisfaction Satisfaction will be evaluated using a 5-point Likert scale, where 1 = not satisfied and 5 = very satisfied, based on verbal feedback from both the patient and the surgeon.

Nausea and Vomiting

Nausea and vomiting will be scored using a 4-point scale:

0 = none

1. = mild
2. = moderate
3. = severe

Potential Complications Any complications associated with the block or the surgical procedure (e.g., hematoma, pneumothorax, local anesthetic toxicity, vascular puncture, or infection) will be recorded.

Length of Hospital Stay The duration from the end of surgery to hospital discharge will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 18-65 years
* American Society of Anesthesiologists (ASA) physical status I-III
* Body Mass Index (BMI) less than 35 kg/m²
* Unilateral breast cancer surgery

Exclusion Criteria:

* Patient refusal to participate
* BMI greater than or equal to 35 kg/m²
* ASA physical status IV-V
* Known allergy to any study medications
* Pregnancy or breastfeeding
* Presence of neuromuscular diseases
* Chronic opioid use
* Chronic pain syndromes
* Significant organ failure (e.g., cardiac, hepatic, renal)
* Contraindications to regional nerve blocks
* Bilateral breast surgery

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2025-05-25 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2026-01-27 (Actual)

PRIMARY OUTCOMES:
Total opioid consumption | the first 24 hours postoperatively
  Total opioid consumption (mg) in the first 24 hours postoperatively, measured using a PCA device.

SECONDARY OUTCOMES:
Postoperative Visual Analog Scale (VAS) Scores - Static and Dynamic Pain | 1, 3, 6, 12, and 24 hours postoperatively.
  Pain intensity will be evaluated using the Visual Analog Scale (VAS) at rest (static) and during movement (dynamic) at postoperative hours 1, 3, 6, 12, and 24. The VAS is scored from 0 (no pain) to 10 (worst imaginable pain), with higher scores indicating worse pain.
Block performance time | During the procedure (from ultrasound probe-skin contact until needle withdrawal, assessed preoperatively)
  Time from ultrasound probe-skin contact to needle withdrawal after injection.
Number of needle passes | During the procedure (number of times the needle trajectory was changed without full withdrawal after skin entry, assessed preoperatively)
  Number of times the needle trajectory was changed after skin entry without full withdrawal.
Quality of recovery assessed by the QoR-15 scale. | 24 hours postoperatively.
  Quality of recovery will be assessed using the QoR-15 scale (range: 0-150), where higher scores indicate better recovery.
Time to first analgesic request. | Within 24 hours postoperatively
  The duration from patient enrollment to the first request for pain relief.
Patient and surgeon satisfaction (5-point Likert scale). | 24 hours postoperatively
  Satisfaction will be assessed using a 5-point Likert scale, ranging from 1 (very dissatisfied) to 5 (very satisfied)
intraoperative opioid consumption | During the surgery(From patient intubation to patient extubation)
  Intraoperative opioids consumption (remifentanyl measured as mcg/kg)

CONTACTS AND LOCATIONS:
Overall Officials: Nilgun Kavrut Ozturk, professor, Study Director — Antalya Training and Research Hospital; Yunus Emre Songur, Resident, Principal Investigator — Antalya Training and Research Hospital; Bahadır Ciftci, Assoc Prof, Principal Investigator — Medipol Mega University Hospital
Locations (1):
- Antalya Training and Research Hospital, Antalya, Turkey (Türkiye)